CLINICAL TRIAL: NCT01632124
Title: Rituximab-induced Pulmonary Function Changes - an Observational Study in Patients With Rheumatoid Arthritis and Inflammatory Myositis
Brief Title: Rituximab-induced Pulmonary Function Changes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: RTX
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Rheumatoid Arthritis; Inflammatory Myositis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Transfer Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Lung function measurement — Spirometry and measurement of diffusing capacity for carbon monoxide
  Other Names: Spirometry; CO diffusing capacity

SUMMARY:
Measuring lung function (FVC, FEV1, DLCO) before, during and after treatment with rituximab in patients with rheumatoid arthritis or inflammatory myositis.

DETAILED DESCRIPTION:
The objective of this study is to investigate whether rituximab (RTX), a drug commonly prescribed in patients with rheumatoid arthritis (RA) or inflammatory myositis, is associated with subclinical interstitial lung disease (ILD). Surrogate markers for interstitial lung diseases are a decrease of the forced vital capacity (FVC) and/or the diffusing capacity of the lung for carbon monoxide (DLCO). However, the measurement of these lung function parameters is indicated as regular follow-up examinations during the treatment with RTX according to the principles of "good clinical practice". We will perform pulmonary function testing (spirometry) including measurement of the DLCO in patients with RA, who are going to be treated with RTX. A baseline lung function measurement will be performed immediately before RTX therapy is started. Follow-up measurements will be performed at 2 weeks, 4 weeks, 8 weeks and 6 months after initiation of RTX therapy. A reduction in forced vital capacity (FVC) of >10% or a fall of >15% in DLCO will be defined as indicative for ILD.

ELIGIBILITY:
Inclusion criteria: - Patients with established diagnosis of RA or inflammatory myositis, in whom a de novo RTX treatment is indicated

* Age >18 y
* Informed consent of patient

Exclusion criteria: - Acute infection

* Pre-existing interstitial pulmonary disease
* Patients with impaired forced vital capacity (FVC) on spirometry (<80% predicted) or with impaired DLCO (<75% predicted).
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients at University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Division of Internal Medicine
Locations (1):
- University Hospital Zurich, Division of Internal Medicine, Zurich, Canton of Zurich, Switzerland